CLINICAL TRIAL: NCT03019536
Title: Multiple-Dose, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY3303560 in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild to Moderate Alzheimer's Disease
Brief Title: A Study of LY3303560 in Participants With Mild Cognitive Impairment or Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16452; I8G-MC-LMDD (Other: Eli Lilly and Company); 2016-002102-39 (EudraCT Number)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 70 mg LY3303560 (Experimental): 70 milligram (mg) LY3303560 administered intravenously (IV) every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to 6 further doses), followed by a 16-week follow-up period.
  Interventions: Drug: LY3303560 - IV; Drug: Placebo - IV; Drug: Florbetapir F 18; Drug: Flortaucipir F18
- 210 mg LY3303560 (Experimental): 210 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to 6 further doses), followed by a 16-week follow-up period.
  Interventions: Drug: LY3303560 - IV; Drug: Placebo - IV; Drug: Florbetapir F 18; Drug: Flortaucipir F18
- Placebo IV (Experimental): Placebo administered intravenously (IV) every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to 6 further doses),, followed by a 16-week follow-up period.
  Interventions: Drug: Placebo - IV; Drug: Florbetapir F 18; Drug: Flortaucipir F18

INTERVENTIONS:
Drug: LY3303560 - IV — Administered IV
  Arms: 210 mg LY3303560; 70 mg LY3303560
Drug: Placebo - IV — Administered IV
Drug: Florbetapir F 18 — Administered IV during the Positron Emission Tomography (PET) scan performed during screening.
Drug: Flortaucipir F18 — Administered IV during the PET scan performed during the study.
  Other Names: AV-1451; [F-18]T807; LY3191748

SUMMARY:
The study involves repeated doses of LY3303560 given by infusion for 49 weeks. The study will examine how safe repeated doses of LY3303560 are, whether they cause side effects in participants with mild cognitive impairment or Alzheimer's Disease, and how LY3303560 is handled by the body and acts in the body. This study will last up to 65 weeks, not including screening. Screening is required within 90 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment (MCI) due to Alzheimer's Disease (AD) or mild-to-moderate AD based on National Institute of Aging and Alzheimer's Association diagnostic criteria
* Female participants: women not of child-bearing potential may participate, and include those who are:

  * Infertile due to surgical sterilisation (hysterectomy, bilateral oophorectomy, or for countries outside of Japan, tubal ligation), congenital anomaly such as mullerian agenesis; or
  * Postmenopausal defined as women at least 50 years of age with an intact uterus who have not taken hormones or oral contraceptives within 1 year, who have had either cessation of menses for at least 1 year, or 6 to 12 months of spontaneous amenorrhea with follicle-stimulating greater than (>) 40 milli-international units per millilitre (mIU/mL)
* Have a body weight of at least 50 kilogram (kg) (except for Japanese sites) and have a body mass index (BMI) of 18.0 to 35.0 kilogram per meter square (kg/m²) (for all sites), inclusive, at screening

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days (3 months and 4 months for sites in the European Union [EU] and Japan, respectively) in a clinical trial involving an IP. If the previous IP has a long half-life, 3 months (4 months for sites in Japan) or 5 half-lives (whichever is longer) should have passed
* Have known allergies to LY3303560, related compounds or any components of the formulation, or history of significant atopy
* Have significant allergies to humanised monoclonal antibodies, diphenhydramine, adrenaline, or methylprednisolone; or have a history of clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Have an increased risk of seizures as evidenced by a history of head trauma with loss of consciousness within the last 5 years or any seizure; prior electroencephalogram with epileptiform activity; surgery to the cerebral cortex; or history within the last 5 years of a serious infectious disease affecting the brain
* Have any contraindications for Magnetic Resonance Imaging (MRI) studies, including claustrophobia, or the presence of metal (ferromagnetic) implants or a cardiac pacemaker
* Have a history of intracranial haemorrhage, cerebrovascular aneurysm, or arteriovenous malformation, carotid artery occlusion, or epilepsy
* Have received acetylcholinesterase inhibitors (AChEIs), memantine, and/or other AD therapy for less than 4 weeks, or have less than 4 weeks of stable therapy on these treatments by time of randomisation (including less than 4 weeks since stopping AChEIs and/or memantine); or have received medications that affect the central nervous system, except treatments for AD, for less than 4 weeks at a stable dose
* Have used stable medical therapy for less than 2 months by time of randomization for any concurrent medical condition that is not exclusionary
* Are currently using or intend to use drugs known to significantly prolong the QT interval, or who have a known risk factor for Torsades de Pointes. A participant will not be excluded if they have been using stable medication that is known to potentially cause significant prolongation of the QT interval, but does not present with any clinically significant prolongation of the QT interval at screening, in the opinion of the investigator
* History of cancer within the last 5 years, with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, non-progressive prostate cancer, or other cancers with low risk of recurrence or spread.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (5):
  - Bioclinica, Melbourne, Florida
  - Bioclinica, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Bioclinica, The Villages, Florida
  - Princeton Medical Institute, Princeton, New Jersey
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kurume
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Bath
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Willis BA, Lo AC, Dage JL, Shcherbinin S, Chinchen L, Andersen SW, LaBell ES, Perahia DGS, Hauck PM, Lowe SL. Safety, Tolerability, and Pharmacokinetics of Zagotenemab in Participants with Symptomatic Alzheimer's Disease: A Phase I Clinical Trial. J Alzheimers Dis Rep. 2023 Sep 15;7(1):1015-1024. doi: 10.3233/ADR-230012. eCollection 2023. PMID 37849628
- See also: Click here for more information about this study: A Study of LY3303560 in Participants With Mild Cognitive Impairment or Alzheimer's Disease — https://trials.lilly.com/en-US/trial/122040

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo IV: Placebo administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to 6 further doses), followed by a 16-week follow-up period.
- 70 mg LY3303560: 70 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to 6 further doses), followed by a 16-week follow-up period.
Period: Overall Study
Arm/Group | Placebo IV | 70 mg LY3303560 | 210 mg LY3303560
Started | 6 | 7 | 9
Received at Least One Dose of Study Drug | 6 | 7 | 9
Completed | 5 | 6 | 7
Not Completed | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo IV: Placebo administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to g further doses), followed by a 16-week follow-up period.
- 70 mg LY3303560: 70 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to g further doses), followed by a 16-week follow-up period.
- 210 mg LY3303560: 210 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up to g further doses), followed by a 16-week follow-up period.
- Total: Total of all reporting groups
Arm/Group | Placebo IV | 70 mg LY3303560 | 210 mg LY3303560 | Total
Number analyzed (Participants) | 6 | 7 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 5 | 6 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 9
  Male | 2 | 6 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 6 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 6 | 14
  Japan | 2 | 1 | 2 | 5
  United Kingdom | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other non-serious adverse events (AEs), and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to Week 65
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo IV: Placebo administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up 6 further doses), followed by a 16-week follow-up period.
- 70 mg LY3303560: 70 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up 6 further doses), followed by a 16-week follow-up period.
- 210 mg LY3303560: 210 mg LY3303560 administered IV every 4 weeks with the option of continuing treatment up to 49 weeks, followed by a 16-week follow-up period.
Arm/Group | Placebo IV | 70 mg LY3303560 | 210 mg LY3303560
Number analyzed (Participants) | 6 | 7 | 9
Participants | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of LY3303560 at Week 49
Description: PK Cmax at Week 49
Time Frame: Week 49 (Pre-dose, 0.5, 2, 4, 8, 336, 672, 1344, 2016, 2688 hours post-dose)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- 210 mg LY3303560: 210 mg LY3303560 administered IV every 4 weeks for 25 weeks with the option of continuing treatment up to 49 weeks (up 6 further doses), followed by a 16-week follow-up period.
Arm/Group | 70 mg LY3303560 | 210 mg LY3303560
Number analyzed (Participants) | 6 | 8
micrograms per milliliter (µg/mL) | 29.2 (23) | 83.9 (22)

3. Secondary Outcome: Pharmacokinetics: Area Under the Serum Concentration Time Curve During the Dosing Interval (AUC 0-tau) of LY3303560
Description: PK: AUC 0-tau at Week 49.
Time Frame: Week 49 (Pre-dose, 0.5, 2, 4, 8, 336, 672, 1344, 2016, 2688 hours post-dose)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (µg*hr/mL)
Arm/Group | 70 mg LY3303560 | 210 mg LY3303560
Number analyzed (Participants) | 5 | 8
microgram*hour per milliliter (µg*hr/mL) | 9140 (21) | 24200 (19)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 65
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo IV | 70 mg LY3303560 | 210 mg LY3303560
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 2/9
Other Adverse Events (participants affected / at risk) | 4/6 | 7/7 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=6) | 70 mg LY3303560 (N=7) | 210 mg LY3303560 (N=9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=6) | 70 mg LY3303560 (N=7) | 210 mg LY3303560 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (8) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urogram (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebellar microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03019536/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03019536/SAP_001.pdf